CLINICAL TRIAL: NCT06419270
Title: Cardiovascular, Renal, and Skeletal Complications in Patients With Post-Surgical Hypoparathyroidism
Acronym: CAREHYPO
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VK-1-10-72-169-23
Record Dates: First submitted 2024-05-07; First posted 2024-05-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-09

CONDITIONS: Hypoparathyroidism; Cardiovascular Complication; Fractures, Bone; Renal Disease
MeSH Terms: conditions — Hypoparathyroidism; Fractures, Bone; Kidney Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples and urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with post-surgical hypoparathyroidism
  Interventions: Other: Observation
- Controls: Gender and age matched controls from the general population
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observational

SUMMARY:
The aim of this observational study is to learn about long term effects to post surgical hypoparathyroidism. The main questions are:

1. Patients with hypoparathyroidism do not have an increased arterial stiffness compared to healthy controls.
2. Patients with hypoparathyroidism do not have an increased coronary artery plaque burden assessed by cardiac CT compared to healthy controls.
3. Patients with hypoparathyroidism do not have an increased prevalence of vertebral fractures compared to healthy controls.

Results will be compared with gender and age matched controls from the general population.

Participants will have a CT scan, DXA scan, tonometry, blood samples and questionaries performed and collect a 24-hour urine sample.

DETAILED DESCRIPTION:
Hypoparathyroidism is a rare endocrine disorder characterized by hypocalcemia with low or undetectable levels of parathyroid hormone. The most common cause of hypoparathyroidism is following neck surgery, whereas approximately 25% of hypoparathyroidism patients are suffering from non-surgical hypoparathyroidism due to e.g., genetic or autoimmune causes. According to updated international guidelines, the condition is considered chronic if treatment with calcium and activated vitamin D is still needed a year after surgery.

A large retrospective cohort study of patients with chronic hypoparathyroidism shows that patients with chronic hypoparathyroidism have a significantly higher risk of cardiovascular disease, compared to patients without hypoparathyroidism. Additionally, it is well known that patients with hypoparathyroidism are at increased risk of renal and extra-skeleton calcifications, although cardiovascular calcifications are only sparsely investigated. Furthermore, both higher arterial stiffness assessed by pulse wave velocity and an increased heart rate have previously been shown in patients with non-surgical hypoparathyroidism. It is largely unknown whether this also applies to patients with post-surgical hypoparathyroidism.

The overall aim of the project is to investigate cardiovascular, renal, and skeletal indices in patients diagnosed with Post Surgical hypoparathyroidism and test the following (null-)hypotheses:

1. H0: Patients with post-surgical hypoparathyroidism do not have an increased arterial stiffness compared to healthy controls.
2. H0: Patients with post-surgical hypoparathyroidism do not have an increased coronary artery plaque burden assessed by cardiac CT compared to healthy controls.
3. H0: Patients with post-surgical hypoparathyroidism do not have an increased prevalence of vertebral fractures compared to healthy controls.

Patients and controls who accept participation will undergo a detailed examination in terms of: Medical history, physical examination, questionnaires, blood and 24-hour urine samples, DXA scan, HRpQCT, tonometry, 12-lead electrocardiogram, 24-hour blood pressure and a CT scan

Data are analyzed according to their distribution using parametric or non-parametric statistics. To address the hypotheses, statistical power calculations have been performed.

50 patients with post-surgical hypoparathyroidism will be matched on sex and age (± 2 years) with 50 randomly selected otherwise healthy controls from the general population.

ELIGIBILITY:
Inclusion Criteria:

Patients only:

* Chronic post surgical hypoparathyroidism diagnosed > 5 years ago. (In case recruitment is too challenging, we will accept duration of disease of minimum one year. Including patients with longest duration of disease first.)
* Require treatment with active vitamin D ≥ 1 µg/day

Controls only:

* No history of neck surgery
* No history of parathyroid disease

All participants:

* Age ≥ 18 years
* 25(OH)D vitamin ≥ 50 nmol/L
* Serum magnesium ≥ 0,50 mmol/L
* Able to read and understand Danish
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m3
* Active cancer or former (except thyroid and basal cell skin) cancer treatment < 5 year ago
* Pregnancy, or breastfeeding < 1 year ago
* Untreated thyroid or liver diseases during the last year
* Treatment with lithium within the last 4 weeks
* Known allergy or sensitivity to iodine
* Any reason that in the opinion of the investigator, that would prevent the patient from completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from endocrine clinics Controls will be recruited from the general population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-05-26 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | 24 months
  aortic pulse wave velocity in m/s
Vertebral fractures | 24 months
  VFA assessing fractures in numbers
coronary artery plaque burden | 24 months
  Heart CT scan assessing coronary artery calcium score

SECONDARY OUTCOMES:
Renal indices | 24 months
  Description of calcifications
bone indices | 24 months
  Description of bone status
Cardiovascular indices | 24 months
  Description of calcifications

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided